CLINICAL TRIAL: NCT01495702
Title: A Phase 3b Randomized, Open Label Study to Evaluate Switching From Regimens Consisting of a Non-nucleoside Reverse Transcriptase Inhibitor (NNRTI) Plus Emtricitabine (FTC) and Tenofovir DF (TDF) to the Elvitegravir/Cobicistat/ Emtricitabine/Tenofovir Disoproxil Fumarate Single-Tablet Regimen (EVG/COBI/FTC/TDF) in Virologically Suppressed, HIV 1 Infected Patients
Brief Title: Study to Evaluate Switching From Regimens Consisting of a Nonnucleoside Reverse Transcriptase Inhibitor Plus Emtricitabine and Tenofovir DF to the Elvitegravir/Cobicistat/Emtricitabine/Tenofovir DF Single-Tablet Regimen in Virologically Suppressed, HIV-1 Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-236-0121; 2011-004963-56 (EudraCT Number)
Record Dates: First submitted 2011-12-14; First posted 2011-12-20 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: HIV-1; HIV; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stribild (Experimental): Participants will switch from their baseline treatment regimen to Stribild for up to 96 weeks, and may continue to receive Stribild in the extension phase.
  Interventions: Drug: Stribild
- NNRTI+FTC/TDF (Active Comparator): Participants will stay on their baseline treatment regimen antiretroviral regimen consisting of an NNRTI plus FTC/TDF for up to 96 weeks, and may switch to Stribild in the extension phase.
  Interventions: Drug: NNRTI; Drug: FTC/TDF; Drug: Stribild

INTERVENTIONS:
Drug: NNRTI — NNRTI agents administered according to prescribing information; allowed NNRTIs include efavirenz (EFV), nevirapine, or rilpivirine.
  Arms: NNRTI+FTC/TDF
Drug: FTC/TDF — FTC/TDF (200/300 mg) administered according to prescribing information
  Other Names: Truvada
  Arms: NNRTI+FTC/TDF
Drug: Stribild — Stribild® (elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate; E/C/F/TDF) (150/150/200/300 mg) STR administered orally once daily with food

SUMMARY:
This study will evaluate the noninferiority of Stribild® (elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (E/C/F/TDF)) single-tablet regimen (STR) relative to regimens consisting of a nonnucleoside reverse transcriptase inhibitor (NNRTI) plus Truvada® (FTC/TDF) in maintaining HIV-1 RNA < 50 copies/mL at Week 48 in virologically suppressed, HIV-1 infected adults. This study will also evaluate the safety, tolerability, and efficacy of the two regimens through 96 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent form
* Be stable on the current formulation(s) of an antiretroviral regimen consisting of an NNRTI plus FTC/TDF for ≥ 6 consecutive months preceding the screening visit. This includes those who began a regimen with individual drug components and subsequently simplified to include a fixed-dose combination formulation of the same drugs.
* Be on the first or second antiretroviral regimen with documented undetectable plasma HIV 1 RNA levels for ≥ 6 months preceding the screening visit
* No previous use of any approved or experimental integrase strand transfer inhibitor (INSTI) for any length of time
* Documented historical genotype prior to starting initial antiretroviral therapy showing no known resistance to TDF or FTC
* HIV RNA < 50 copies/mL at screening
* Normal ECG
* Hepatic transaminases ≤ 5 × the upper limit of the normal range (ULN)
* Total bilirubin ≤ 1.5 mg/dL
* Adequate hematologic function
* Serum amylase ≤ 5 × ULN
* Estimated glomerular filtration rate ≥ 70 mL/min
* Females of childbearing potential must agree to utilize protocol recommended contraception methods or be nonheterosexually active, practice sexual abstinence from screening throughout the duration of the study period and for 12 weeks for participants on EFV/FTC/TDF or efavirenz or 30 days for the rest of participants following the last dose of study drug
* Female participants who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing
* Male participants must agree to utilize protocol-recommended methods of contraception during heterosexual intercourse or be nonheterosexually active, and practice sexual abstinence from the screening visit.
* Age ≥ 18 years

Exclusion Criteria:

* New AIDS-defining condition diagnosed within the 30 days prior to screening
* Females who are breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Receiving drug treatment for hepatitis C, or those who are anticipated to receive treatment for hepatitis C during the course of the study
* Experiencing decompensated cirrhosis
* Have an implanted defibrillator or pacemaker
* Current alcohol or substance abuse that would interfere with compliance
* A history of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma (KS), basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma. Persons with cutaneous KS are eligible, but must not have received any systemic therapy for KS within 30 days of baseline and must not be anticipated to require systemic therapy during the study.
* Active, serious infections requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Have been treated with immunosuppressant therapies or chemotherapeutic agents within 3 months of study screening, or expected to receive these agents or systemic steroids during the study
* Receiving ongoing therapy with any of the medications, including drugs not to be used with elvitegravir, cobicistat, FTC, or TDF; or those with any known allergies to the excipients of E/C/F/TDF tablets, or FTC/TDF tablets
* No anticipated need to initiate drugs during the study that are contraindicated
* Receiving other investigational drugs
* Participation in any other clinical trial
* Any other clinical condition or prior therapy that would make the participant unsuitable for the study or unable to comply with the dosing requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damian McColl, Study Director — Gilead Sciences
Locations (80):
- United States (39):
  - Spectrum Medical Group, Phoenix, Arizona
  - AHF Research Center, Beverly Hills, California
  - Pacific Oak Medical Group, Beverly Hills, California
  - Kaiser Permanente, Hayward, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - OASIS Clinic, Los Angeles, California
  - Anthony Mills MD Inc, Los Angeles, California
  - Alameda County Medical Center, Oakland, California
  - Kaiser Permanente Medical Group, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Metropolis Medical, San Francisco, California
  - Kaiser Permanente, San Francisco, California
  - Dupont Circle Physicians Group, P.C., Washington D.C., District of Columbia
  - Capital Medical Associates, P.C., Washington D.C., District of Columbia
  - Gary Richmond MD, PA, Inc, Fort Lauderdale, Florida
  - Midway Immunology and Research, Ft. Pierce, Florida
  - The Kinder Medical Group, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - ValuHealth MD, LLC, Orlando, Florida
  - Infectious Diseases Associates of Northwest Florida, Pensacola, Florida
  - Health Positive, Safety Harbor, Florida
  - Atlanta ID Group, PC, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Be Well Medical Center, Berkley, Michigan
  - HIV Program Hennepin County Medical Center, Minneapolis, Minnesota
  - The Kansas City Free Health Clinic, Kansas City, Missouri
  - ID Care, Hillsborough, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Greiger Clinic, Mount Vernon, New York
  - Aaron Diamond AIDS Research Center, New York, New York
  - ID Consultants, P.A., Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Southwest Infectious Disease Clinical Researach Inc, Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Therapeutic Concepts PA, Houston, Texas
  - Gordon E. Crofoot MD, PA, Houston, Texas
  - Clinical Alliance for Research & Education - Infectious Disease, Annandale, Virginia
- Australia (3):
  - Holdsworth House Medical Practice, Darlinghurst
  - Prahran Market Clinic, South Yarra
  - East Sydney Doctors, Sydney
- Austria (2):
  - Medical University of Vienna, Vienna
  - Otto Wagner Spital, Vienna
- Belgium (3):
  - SEAMEO Regional Centre for Tropical Medicine, Antwerp
  - Hôpitaux IRIS Sud, Brussels
  - University Hospital of Leuven, Leuven
- Canada (3):
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Maple Leaf Medical Clinic, Toronto, Ontario
  - Clinique Medicale Du Quartier Latin, Montreal, Quebec
- France (5):
  - CHU de Besancon - Hopital Saint-Jacques, Besançon
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Hopital Saint Louis, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Hopital Saint Antoine, Paris
- Germany (7):
  - EPIMED GmbH, Berlin
  - MIB Dienstleistung GmbH, Berlin
  - Medizinische Universitätsklinik, Bonn
  - Infektiologikum, Frankfurt
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - ICH Study Center, Hamburg
  - MUC Research GmbH, München
- Italy (5):
  - Azienda Ospedaliera Ospedale di Circolo Busto Arsizio, Busto Arsizio/Varese
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Ospedale Luigi Sacco, Milan
  - Istituto Nazionale Malattie Infettive "Lazzaro Spallanzani" IRCCS, Roma
  - Policlinico Universitario Agostino Gemelli, Rome
- Hospital de Santa Maria - CHLN EPE, Lisbon, Portugal
- Clinical Research Puerto Rico Inc, San Juan, Puerto Rica, Puerto Rico
- Spain (5):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital del Mar, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital La Fe de Valencia, Valencia
- United Kingdom (6):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Western General Hospital, Edinburgh
  - Homerton University Hospital, London
  - South London Healthcare NHS Trust, London
  - St. Thomas' Hospital, London
  - Chelsea & Westminster Hospital, London

REFERENCES:
- [Derived] Pozniak A, Flamm J, Antinori A, Bloch M, Ward D, Berenguer J, Cote P, Andreatta K, Garner W, Szwarcberg J, Nguyen-Cleary T, McColl DJ, Piontkowsky D. Switching to the single-tablet regimen of elvitegravir, cobicistat, emtricitabine, and tenofovir DF from non-nucleoside reverse transcriptase inhibitor plus coformulated emtricitabine and tenofovir DF regimens: Week 96 results of STRATEGY-NNRTI. HIV Clin Trials. 2017 Jul;18(4):141-148. doi: 10.1080/15284336.2017.1338844. Epub 2017 Jul 9. PMID 28689453
- [Derived] Pozniak A, Markowitz M, Mills A, Stellbrink HJ, Antela A, Domingo P, Girard PM, Henry K, Nguyen T, Piontkowsky D, Garner W, White K, Guyer B. Switching to coformulated elvitegravir, cobicistat, emtricitabine, and tenofovir versus continuation of non-nucleoside reverse transcriptase inhibitor with emtricitabine and tenofovir in virologically suppressed adults with HIV (STRATEGY-NNRTI): 48 week results of a randomised, open-label, phase 3b non-inferiority trial. Lancet Infect Dis. 2014 Jul;14(7):590-9. doi: 10.1016/S1473-3099(14)70796-0. Epub 2014 Jun 5. PMID 24908550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, and Australia. The first participant was screened on 13 December 2011. The last study visit occurred on 01 December 2014.
Pre-assignment Details: 571 participants were screened.
Groups:
- Stribild: Participants switched from their baseline treatment regimen to Stribild® (elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate; E/C/F/TDF) (150/150/200/300 mg) single-tablet regimen (STR) once daily for up to 96 weeks in the randomized phase, and may have continued to receive Stribild in the extension phase.
- NNRTI+FTC/TDF: Participants stayed on their baseline treatment regimen consisting of an nonnucleoside reverse transcriptase inhibitor (NNRTI) (efavirenz (EFV), nevirapine (NVP), or rilpivirine (RPV)) plus emtricitabine (FTC)/TDF (200/300 mg) (administered according to prescribing information) for up to 96 weeks in the randomized phase, and may have switched to Stribild in the extension phase.
Period: Randomized Phase
Arm/Group | Stribild | NNRTI+FTC/TDF
Started | 292 | 147
Completed | 266 | 119
Not Completed | 26 | 28
Not completed — Randomized But Not Treated | 1 | 4
Not completed — Adverse Event | 2 | 2
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Investigators Discretion | 2 | 0
Not completed — Withdrew Consent | 10 | 18
Not completed — Lost to Follow-up | 4 | 3
Not completed — Participant Noncompliance | 1 | 0
Not completed — Protocol Violation | 3 | 1
Period: Extension Phase
Arm/Group | Stribild | NNRTI+FTC/TDF
Started | 26 | 2
Completed | 26 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants were randomized and received at least one dose of study drug
Groups:
- Stribild: Participants switched from their baseline treatment regimen to Stribild (E/C/F/TDF) (150/150/200/300 mg) STR once daily for up to 96 weeks in the randomized phase, and may have continued to receive Stribild in the extension phase.
- NNRTI+FTC/TDF: Participants stayed on their baseline treatment regimen consisting of an NNRTI (EFV, NVP, or RPV) plus FTC/TDF (200/300 mg) (administered according to prescribing information) for up to 96 weeks in the randomized phase, and may have switched to Stribild in the extension phase.
- Total: Total of all reporting groups
Arm/Group | Stribild | NNRTI+FTC/TDF | Total
Number analyzed (Participants) | 291 | 143 | 434
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (9.6) | 40 (9.7) | 41 (9.7)
Age, Customized [Number; unit: participants]
  < 40 years | 114 | 74 | 188
  ≥ 40 to < 50 years | 106 | 44 | 150
  ≥ 50 years | 71 | 25 | 96
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 9 | 32
  Male | 268 | 134 | 402
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 4 | 9 | 13
  Black or African Heritage | 49 | 23 | 72
  Native Hawaiian or Pacific Islander | 1 | 0 | 1
  White | 231 | 109 | 340
  Other | 4 | 2 | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 30 | 16 | 46
  Non-Hispanic/Latino | 261 | 127 | 388
  Not Permitted | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 4 | 1 | 5
  Portugal | 2 | 4 | 6
  United States | 152 | 75 | 227
  Puerto Rico | 4 | 2 | 6
  Canada | 13 | 6 | 19
  Spain | 27 | 13 | 40
  Belgium | 14 | 7 | 21
  Austria | 6 | 3 | 9
  Australia | 8 | 4 | 12
  Germany | 24 | 10 | 34
  United Kingdom | 13 | 5 | 18
  Italy | 24 | 13 | 37
HIV-1 RNA Category [Number; unit: participants]
  < 50 copies/mL | 285 | 141 | 426
  50 to < 200 copies/mL | 4 | 2 | 6
  200 to < 400 copies/mL | 0 | 0 | 0
  ≥ 400 copies/mL | 2 | 0 | 2
CD4+ Cell Count [Mean (Standard Deviation); unit: cells/µL] | 586 (210.3) | 593 (224.6) | 588 (214.9)
CD4+ Cell Count Category [Number; unit: participants]
  ≤ 50 cells/µL | 0 | 0 | 0
  51 to ≤ 200 cells/µL | 4 | 1 | 5
  201 to ≤ 350 cells/µL | 26 | 20 | 46
  351 to ≤ 500 cells/µL | 75 | 33 | 108
  > 500 cells/µL | 186 | 89 | 275
HIV Disease Status [Number; unit: participants]
  Asymptomatic | 225 | 115 | 340
  Symptomatic HIV Infections | 36 | 14 | 50
  AIDS | 30 | 14 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48
Description: The FDA-defined Snapshot algorithm was used, which defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time.
Time Frame: Week 48
Population: Full Analysis Set: participants were randomized, received at least 1 dose of study drug, had no documented resistance, and were on an NNRTI at screening
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | NNRTI+FTC/TDF
Number analyzed (Participants) | 290 | 143
percentage of participants | 93.4 | 88.1
Statistical Analysis 1: Comparison: Stribild vs NNRTI+FTC/TDF; Test type: Non-Inferiority or Equivalence — The null hypothesis was that the Stribild group was at least 12% worse than the NNRTI+FTC/TDF group with respect to the percentage of participants maintaining HIV-1 RNA < 50 copies/mL at Week 48. The alternative hypothesis was that the Stribild group was less than 12% worse than the NNRTI+FTC/TDF group; p = 0.066, Fisher Exact; Difference in proportions = 5.3, 95% CI 2-sided [-0.5 to 12.0] — The 95% confidence interval (CI) for the difference was from unconditional exact method using 2 inverted 1-sided tests with the standardized statistic using StatXact

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96
Description: as for outcome 1
Time Frame: Week 96
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | NNRTI+FTC/TDF
Number analyzed (Participants) | 290 | 143
percentage of participants | 86.6 | 80.4

3. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed; the missing-equals-excluded approach where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Stribild | NNRTI+FTC/TDF
Number analyzed (Participants) | 270 | 126
cells/µL | 56 (147.3) | 58 (179.3)

4. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 96
Time Frame: Baseline; Week 96
Population: Participants in the Full Analysis Set with available data while on study drug were analyzed; the missing-equals-excluded approach where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Stribild | NNRTI+FTC/TDF
Number analyzed (Participants) | 256 | 116
cells/µL | 83 (166.7) | 101 (156.5)

ADVERSE EVENTS:
Time Frame: Baseline through end of study (average 90 weeks)
Description: Safety Analysis Set participants were randomized and received at least 1 dose of study drug
Groups:
- Stribild (Randomized Phase): Adverse events for this reporting group include those occurring in participants receiving Stribild in the randomized phase.
  Participants switched from their baseline treatment regimen to Stribild (E/C/F/TDF) (150/150/200/300 mg) STR once daily for up to 96 weeks in the randomized phase, and may have continued to receive Stribild in the extension phase.
- NNRTI+FTC/TDF (Randomized Phase): Adverse events for this reporting group include those occurring in participants receiving NNRTI+FTC/TDF in the randomized phase.
  Participants stayed on their baseline treatment regimen consisting of an NNRTI (EFV, NVP, or RPV) plus FTC/TDF (200/300 mg) (administered according to prescribing information) for up to 96 weeks in the randomized phase, and may have switched to Stribild in the extension phase.
- All Stribild: Adverse events for this reporting group include those occurring in all participants while receiving Stribild in the randomized and extension phases.
Arm/Group | Stribild (Randomized Phase) | NNRTI+FTC/TDF (Randomized Phase) | All Stribild
Serious Adverse Events (participants affected / at risk) | 24/291 | 7/143 | 26/293
Other Adverse Events (participants affected / at risk) | 154/291 | 66/143 | 154/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stribild (Randomized Phase) (N=291) | NNRTI+FTC/TDF (Randomized Phase) (N=143) | All Stribild (N=293)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 1 | 1 | 1
Shigella infection (Infections and infestations) | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 1
Delusion (Psychiatric disorders) | 1 | 0 | 1
Drug abuse (Psychiatric disorders) | 1 | 0 | 1
Stress (Psychiatric disorders) | 1 | 0 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stribild (Randomized Phase) (N=291) | NNRTI+FTC/TDF (Randomized Phase) (N=143) | All Stribild (N=293)
Diarrhoea (Gastrointestinal disorders) | 30 | 11 | 30
Nausea (Gastrointestinal disorders) | 24 | 4 | 24
Fatigue (General disorders) | 19 | 2 | 19
Nasopharyngitis (Infections and infestations) | 30 | 17 | 30
Sinusitis (Infections and infestations) | 21 | 5 | 21
Syphilis (Infections and infestations) | 17 | 10 | 17
Upper respiratory tract infection (Infections and infestations) | 33 | 15 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 5 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 8 | 23
Headache (Nervous system disorders) | 29 | 8 | 29
Insomnia (Psychiatric disorders) | 22 | 11 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 5 | 24

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years